CLINICAL TRIAL: NCT05457478
Title: Evaluation of the Use of "Smart" Body-Weight Scales in Patients With Head and Neck Cancer Undergoing Radiation Therapy
Brief Title: The Use of "Smart" Body-Weight Scales for Weight and Nutritional Monitoring in Patients With Head and Neck Cancer Undergoing Radiation Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI departure
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Cambia Health Foundation (Other); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Ravi Chandra, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00022914; NCI-2022-05054 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00022914 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2022-07-01; First posted 2022-07-14 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Malignant Head and Neck Neoplasm
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 2 (no weighing) (Active Comparator): Patients do not weigh themselves using the "Smart" scale during standard radiation therapy.
  Interventions: Other: Questionnaire Administration
- Cohort I ('Smart" scale weighing) (Experimental): Patients weigh themselves daily using the "Smart" scale over 5-8 weeks during standard radiation therapy.
  Interventions: Other: Medical Device Qardio® smart scale Usage and Evaluation; Other: Questionnaire Administration

INTERVENTIONS:
Other: Medical Device Qardio® smart scale Usage and Evaluation — Weight monitored using a Qardio® smart scale
  Other Names: Smart body-weight scale
  Arms: Cohort I ('Smart" scale weighing)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial studies the use of "smart" body-weight scales to monitor weight and nutrition among patients with head and neck cancer undergoing radiation therapy. Malnutrition affects 30-50% of patients diagnosed with head and neck cancer, and approximately 30% of patients have malnutrition prior to diagnosis. "Smart" body weight scales can possibly make self-weighing easier, faster, and more accurate through weight recordings through mobile applications available for "smart" scales. This has the potential to maximize nutritional guidance through quick weight updates, possibly delaying or removing the use of patient enteral feeding (tube feeding). By avoiding or minimizing the use of enteral feeding during radiation therapy, the risk of long-term tube dependence and swallowing ability complications may be reduced.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the feasibility of "smart" body scales in patients undergoing radiation therapy for head and neck cancer.

SECONDARY OBJECTIVE:

I. MD Anderson Symptom Inventory for Head and Neck Cancer (MDASI-HN) questionnaire, overall pain scores, and weight loss percentage.

OUTLINE: Patients are assigned to 1 of 2 cohorts.

COHORT I: Patients weigh themselves daily using the "Smart" scale over 5-8 weeks during standard radiation therapy.

COHORT II: Patients do not weigh themselves using the "Smart" scale during standard radiation therapy.

After completion of study intervention, patients are followed up within 2 weeks and 3 months post-radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a histologically confirmed malignancy whereby pursual of radiation therapy has potential curative benefits for the patient.
* Criteria for selection of head and neck malignancies include squamous cell carcinoma.
* Ability to understand and the willingness to sign a written informed consent document.
* For the intervention group, the ability to properly utilize a "smart" body weight scale after appropriate training has been provided. This includes access to wireless internet which can be paired with the "smart" body weight scale to transmit weight scale data.

Exclusion Criteria:

* Do not meet the criteria for histologically confirmed malignancies.
* Refuse or do not pursue radiation therapy for curative benefit of their malignancy.
* Who do not understand or are unwilling to sign a written informed consent document.
* For the intervention group, the inability to utilize or pair their "smart" body weight sales to wireless internet.
* Members of vulnerable populations as below
* Pregnant women, children, prisoners, neonates, and decisionally impaired adults will not be included in this study. Excluding vulnerable populations, all patients who are receiving or seeking medical care at Oregon Health & Science University (OHSU) for their head and neck cancer and meet inclusion criteria will be invited to participate in this study. Potential participants will be approached by a member of the clinic staff and will be asked to review a copy of the informed consent form prior to being seen by a treating physician. The investigator, or other qualified, designated healthcare provider will review the informed consent form with potential participants and address any questions or concerns prior to obtaining written informed consent for participation in this study. The investigator or other qualified, designated healthcare provider will also address any future questions or concerns of the participant.

  * Only individuals who have provided directly their written informed consent for participation in this study and meet inclusion criteria will be placed in the study. The participation of patients who are mentally incapacitated (e.g., comatose, unresponsive) will not be sought

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2023-01-13 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-09-13 (Actual)

PRIMARY OUTCOMES:
Adherence to treatment | Up to 8 weeks
  Will include continuous variables (number of times participant stepped on the scale). Standard statistical methods will be utilized to analyze cohort data, while also accounting for missing unused, or spurious data.

SECONDARY OUTCOMES:
MD Anderson Symptom Inventory for Head and Neck Cancer (MDASI-HN) questionnaire scores | Baseline up to 3 months post-radiation therapy
  The MDASI-HN has 13 core symptoms that is scored, at their worst over the last 24 hours, on a 0-10 numeric rating scale. A "0" means that a symptom is not present and a "10" is "as bad as you can imagine." Standard statistical methods will be utilized to analyze cohort data, while also accounting for missing unused, or spurious data.
Overall pain scores | Up to 3 months post-radiation therapy
  Pain scores will be on a numeric rating scale, with lower numbers indicating lower pain values. Standard statistical methods will be utilized to analyze cohort data, while also accounting for missing unused, or spurious data.
Weight loss percentage | Up to 3 months post-radiation therapy
  Standard statistical methods will be utilized to analyze cohort data, while also accounting for missing unused, or spurious data.

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Chandra, Principal Investigator — OHSU Knight Cancer Institute
Locations (2):
- United States (2):
  - Mid-Atlantic Permanente Medical Group, Rockville, Maryland
  - OHSU Knight Cancer Institute, Portland, Oregon